CLINICAL TRIAL: NCT02472769
Title: A Randomized, Double Blind, Parallel-group, Dose Escalation Placebo-controlled Multicenter Study to Investigate the Safety and Tolerability of IBP-9414 Administered in Preterm Infants.
Brief Title: IBP-9414 for the Prevention of Necrotizing Enterocolitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Infant Bacterial Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IBP-9414-010
Record Dates: First submitted 2015-06-02; First posted 2015-06-16 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-01

CONDITIONS: Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- IBP-9414 (Active Comparator): IBP-9414 Oral Daily
  Interventions: Drug: IBP-9414
- Placebo (Placebo Comparator): Sterile water
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IBP-9414
  Arms: IBP-9414
Drug: Placebo — Sterile water
  Arms: Placebo

SUMMARY:
Two different dose levels will be evaluated in two different birth weight categories, compared to placebo with regards to safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age ≤32 weeks
2. Birth weight: a) ≤ 2,000 g and b) ≤ 1,000 g.
3. < 48 hours of age.
4. Written informed consent from the patient's legally authorized representative(s).

Exclusion Criteria:

1. Participation in an additional interventional clinical trial in which an investigational drug will be administered.
2. Infants in extremis to whom no further intensive care is offered by attending neonatologist (e.g., infant being provided only hospice/comfort care).
3. Congenital or acquired gastrointestinal pathology.
4. Other conditions of the infant, which in the opinion of the attending neonatologist, preclude participation.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of IBP-9414 as the observed number of adverse events (AE) and serious adverse events (SAE) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Josef Neu, MD, Principal Investigator — University of Florida College of Medicine, Gainsville, FL
Locations (15):
- United States (15):
  - Univ. Arkansas Medical Sciences, Little Rock, Arkansas
  - UCLA Medical Center, Los Angeles, California
  - University Florida Health, Gainesville, Florida
  - Wolfson Children´s Hospital, Jacksonville, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Wesley Medical Center, Wichita, Kansas
  - Kings County Hospital Center, Brooklyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center of Philadelphia, Philadelphia, Pennsylvania
  - Jackson Madison County General Hospital, Jackson, Tennessee
  - Timpanogos Regional Hospital, Orem, Utah